CLINICAL TRIAL: NCT07111845
Title: Human Doctors or AI: Evaluating Patient Satisfaction in Urinary Stone Disease Consultations
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abant Izzet Baysal University (Other)
Responsible Party: Principal Investigator, H. Alperen YILDIZ, Assistant Professor, Abant Izzet Baysal University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 20243209
Record Dates: First submitted 2025-07-25; First posted 2025-08-08 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-08

CONDITIONS: Patient Satisfaction
Keywords: AI in healthcare; chatbot consultations; patient experience; urinary stone disease; digital medicine
MeSH Terms: conditions — Patient Satisfaction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Doctors Group (Experimental): Participants consult a real urologist.
  Interventions: Behavioral: Medical Consultation
- ChatGPT Group (Experimental): Participants ask all questions to ChatGPT.
  Interventions: Behavioral: Medical Consultation
- Gemini Group (Experimental): Participants ask all questions to Gemini.
  Interventions: Behavioral: Medical Consultation
- Perplexity Group (Experimental): Participants ask all questions to Perplexity.
  Interventions: Behavioral: Medical Consultation
- Copilot Group (Experimental): Participants ask all questions to Microsoft Copilot.
  Interventions: Behavioral: Medical Consultation

INTERVENTIONS:
Behavioral: Medical Consultation — Participants will be randomly assigned to receive medical consultation about urinary stone disease from one of five sources: a real urologist (in-person) or one of four AI chatbots (ChatGPT, Gemini, Perplexity, or Microsoft Copilot). Each participant will be instructed to ask all their questions related to urinary stone disease and continue the consultation until they feel adequately informed. The consultation format (human vs. AI) will depend on group assignment. After the session, participants will complete a validated satisfaction questionnaire (CSQ-8) to assess their experience.

SUMMARY:
The goal of this observational study is to understand how satisfied patients are after getting medical advice about urinary stone disease from either a real doctor or an artificial intelligence (AI) chatbot. We want to learn whether people feel more satisfied with the information and support they get from human doctors or from AI tools like ChatGPT, Gemini, Perplexity, or Copilot.

The main questions it aims to answer are:

* Are patients more satisfied after consulting a real doctor or an AI chatbot?
* Does the time spent in the consultation affect satisfaction?

Researchers will compare doctor consultations with consultations from different AI chatbots to see if there are differences in patient satisfaction.

Participants will:

* Ask all their medical questions about urinary stones to one of the sources (a doctor or a specific AI chatbot)
* Fill out a short questionnaire (CSQ-8) to rate how satisfied they felt with the answers they received

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed with urinary stone disease,
* Aged 18 years or older,
* Provided written informed consent to participate in the study.

Exclusion Criteria:

* History of previous urinary stone disease, stone-related procedures,
* Presence of other acute medical conditions unrelated to urinary stone disease,
* Cognitive or communication impairments,
* Pregnancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2025-01-01 (Actual); Primary Completion 2025-05-20 (Actual); Study Completion 2025-05-30 (Actual)

PRIMARY OUTCOMES:
Patient Satisfaction Score | Within 1 hour after the consultation
  Patient satisfaction will be measured using the validated Client Satisfaction Questionnaire (CSQ-8), which consists of 8 items scored on a 4-point Likert scale. The total score ranges from 8 to 32, with higher scores indicating greater satisfaction.

SECONDARY OUTCOMES:
Consultation Duration | During consultation
  Total duration (in minutes) of the consultation session (doctor or chatbot) will be recorded and compared across all groups.

CONTACTS AND LOCATIONS:
Locations (1):
- İzzet Baysal Eğitim ve Araştırma Hastanesi, Bolu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
The data generated and analysed during the current study are not publicly available due to ethical and privacy concerns but are available from the corresponding author on reasonable request.

REFERENCES:
- [Result] Whiles BB, Bird VG, Canales BK, DiBianco JM, Terry RS. Caution! AI Bot Has Entered the Patient Chat: ChatGPT Has Limitations in Providing Accurate Urologic Healthcare Advice. Urology. 2023 Oct;180:278-284. doi: 10.1016/j.urology.2023.07.010. Epub 2023 Jul 17. PMID 37467806
- [Result] Hanci V, Ergun B, Gul S, Uzun O, Erdemir I, Hanci FB. Assessment of readability, reliability, and quality of ChatGPT(R), BARD(R), Gemini(R), Copilot(R), Perplexity(R) responses on palliative care. Medicine (Baltimore). 2024 Aug 16;103(33):e39305. doi: 10.1097/MD.0000000000039305. PMID 39151545
- [Result] Simon BD, Gelikman DG, Turkbey B. Evaluating the efficacy of artificial intelligence chatbots in urological health: insights for urologists on patient interactions with large language models. Transl Androl Urol. 2024 May 31;13(5):879-883. doi: 10.21037/tau-23-635. Epub 2024 May 7. No abstract available. PMID 38855603

DOCUMENTS (2):
  • Study Protocol (2025-08-01): https://cdn.clinicaltrials.gov/large-docs/45/NCT07111845/Prot_000.pdf
  • Statistical Analysis Plan (2025-08-01): https://cdn.clinicaltrials.gov/large-docs/45/NCT07111845/SAP_001.pdf